CLINICAL TRIAL: NCT02153710
Title: A Prospective, Controlled Study of Rehabilitation of Anomia in Aphasia
Brief Title: Speech Therapy for Aphasia: Comparing Two Treatments
Acronym: PMvSFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Portland State University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O1183-R
Record Dates: First submitted 2014-03-20; First posted 2014-06-03 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Stroke
Keywords: Aphasia; Anomia
MeSH Terms: conditions — Stroke; Aphasia; Anomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phonomotor therapy (Experimental): Experimental group
  Interventions: Behavioral: Phonomotor Therapy
- Semantic Feature Analysis therapy (Active Comparator): Current standard of care therapy
  Interventions: Behavioral: Semantic Feature Analysis therapy

INTERVENTIONS:
Behavioral: Semantic Feature Analysis therapy — Control therapy; current standard of care therapy
  Arms: Semantic Feature Analysis therapy
Behavioral: Phonomotor Therapy — Experimental therapy.
  Arms: Phonomotor therapy

SUMMARY:
This is a behavioral speech therapy trial for individuals who have suffered a stroke on the left side of the brain and have difficulty speaking. The name of this disorder is called "aphasia." Individuals in this study will receive one of two treatments. The first is a phonological (sound level) treatment and the second is a semantic (word level) treatment. Individuals in both groups will receive 60 hours of therapy for free (2 hours/day, 5 days/week, 6 weeks).

DETAILED DESCRIPTION:
Purpose: The ultimate goal of anomia treatment should be to achieve gains in exemplars trained in the therapy session as well as generalization to untrained exemplars and contexts. Phonomotor treatment (PMT) has shown such effects but has not yet been compared to a commonly used lexical/semantic based treatment (semantic feature analysis; SFA).

Methods: In a between group randomized controlled trial, 58 persons with aphasia characterized by anomia and phonological dysfunction were randomized to receive 56-60 hours of intensively delivered treatment over 6 weeks with testing pre-, post- and three-months post treatment termination.

ELIGIBILITY:
Inclusion Criteria:

* Single, left-hemisphere stroke
* English as primary language prior to stroke

Exclusion Criteria:

* Other neurological disorders
* Untreated depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane L. Kendall, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phonomotor Therapy | Semantic Feature Analysis Therapy
Started | 28 | 30
Completed | 28 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Race information was not collected in this study
Groups:
- Total: Total of all reporting groups
Arm/Group | Phonomotor Therapy | Semantic Feature Analysis Therapy | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.6) | 63.4 (12.3) | 63.35 (.070)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 15 | 18 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race was not collected from participants.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Spoken Word Production (Confrontation Naming)
Description: Reporting a change in percent correct scores pre-treatment versus 3-months post treatment. (0-100% scale)
Time Frame: Pretreatment to 3 months following treatment termination change
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Phonomotor Therapy | Semantic Feature Analysis Therapy
Number analyzed (Participants) | 28 | 30
percent correct | 53.01 (29.71) | 50.37 (29.79)

2. Secondary Outcome: Response Latency
Description: Change in response latency of confrontation naming pre-treatment versus 3 months post treatment.
Time Frame: Pretreatment to 3 months following treatment termination change
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Phonomotor Therapy | Semantic Feature Analysis Therapy
Number analyzed (Participants) | 28 | 30
seconds | 1.49 (0.54) | 1.40 (0.67)

3. Secondary Outcome: Verbs Correctly Named
Description: Change in confrontation naming of verbs were scored for accuracy and percent correct (0% to 100%) was analyzed before versus 3 months post treatment.
Time Frame: Pretreatment to 3 months following treatment termination change
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Phonomotor Therapy | Semantic Feature Analysis Therapy
Number analyzed (Participants) | 28 | 30
percent correct | 3.36 (7.19) | 2.46 (9.11)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Phonomotor Therapy | Semantic Feature Analysis Therapy
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2013-10-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT02153710/Prot_000.pdf
  • Informed Consent Form: University of Washington informed consent (2015-03-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT02153710/ICF_001.pdf
  • Informed Consent Form: VA informed consent (2015-05-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT02153710/ICF_002.pdf